CLINICAL TRIAL: NCT01093794
Title: A Bioequivalence Study With Two Tablet Strengths of the Final Market Image (FMI) Sitagliptin/Metformin Fixed Dose Combination (FDC) Tablet
Brief Title: Bioequivalence Study of Sitagliptin/Metformin Combination Tablet (MK0431A-122)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0431A-122; 2010_518
Record Dates: First submitted 2010-03-19; First posted 2010-03-26 (Estimated); Results first posted 2011-06-27 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1. Sit + Met500 / SitMet500 FDC / SitMet850 FDC / Sit + Met850 (Experimental): Participants were administered treatment in the following sequence with a minimum 7 day washout period between treatments:
  * Co-administration of 50 mg sitagliptin and 500 mg metformin
  * sitagliptin/metformin 50 mg/500 mg FDC tablet
  * sitagliptin/metformin 50 mg/850 mg FDC tablet
  * Co-administration of 50 mg sitagliptin and 850 mg metformin
  Interventions: Drug: Co-administration of 50 mg sitagliptin and 500 mg metformin; Drug: sitagliptin/metformin 50 mg/500 mg tablet; Drug: Co-administration of 50 mg sitagliptin and 850 mg metformin; Drug: sitagliptin/metformin 50 mg/850 mg tablet
- 2. SitMet500 FDC / Sit + Met850 / Sit + Met500 / SitMet850 FDC (Experimental): Participants were administered treatment in the following sequence with a minimum 7 day washout period between treatments:
  * sitagliptin/metformin 50 mg/500 mg FDC tablet
  * Co-administration of 50 mg sitagliptin and 850 mg metformin
  * Co-administration of 50 mg sitagliptin and 500mg metformin
  * sitagliptin/metformin 50 mg/850 mg FDC tablet
  Interventions: Drug: Co-administration of 50 mg sitagliptin and 500 mg metformin; Drug: sitagliptin/metformin 50 mg/500 mg tablet; Drug: Co-administration of 50 mg sitagliptin and 850 mg metformin; Drug: sitagliptin/metformin 50 mg/850 mg tablet
- 3. Sit + Met850 / SitMet850 FDC / SitMet500 FDC / Sit + Met500 (Experimental): Participants were administered treatment in the following sequence with a minimum 7 day washout period between treatments:
  * Co-administration of 50 mg sitagliptin and 850 mg metformin
  * sitagliptin/metformin 50 mg/850 mg FDC tablet
  * sitagliptin/metformin 50 mg/500 mg FDC tablet
  * Co-administration of 50 mg sitagliptin and 500mg metformin
  Interventions: Drug: Co-administration of 50 mg sitagliptin and 500 mg metformin; Drug: sitagliptin/metformin 50 mg/500 mg tablet; Drug: Co-administration of 50 mg sitagliptin and 850 mg metformin; Drug: sitagliptin/metformin 50 mg/850 mg tablet
- 4. SitMet850 FDC / Sit + Met500 / Sit + Met850 / SitMet500 FDC (Experimental): Participants were administered treatment in the following sequence with a minimum 7 day washout period between treatments:
  * sitagliptin/metformin 50 mg/850 mg FDC tablet
  * Co-administration of 50 mg sitagliptin and 500 mg metformin
  * Co-administration of 50 mg sitagliptin and 850 mg metformin
  * sitagliptin/metformin 50 mg/500 mg FDC tablet
  Interventions: Drug: Co-administration of 50 mg sitagliptin and 500 mg metformin; Drug: sitagliptin/metformin 50 mg/500 mg tablet; Drug: Co-administration of 50 mg sitagliptin and 850 mg metformin; Drug: sitagliptin/metformin 50 mg/850 mg tablet

INTERVENTIONS:
Drug: Co-administration of 50 mg sitagliptin and 500 mg metformin — Co-administration of 50 mg sitagliptin and 500 mg China-sourced metformin as individual tablets with 240 ml water on Day 1 of the relevant treatment period (Sit + Met500) after fasting for at least 10 hours.
Drug: sitagliptin/metformin 50 mg/500 mg tablet — Single dose administration of the final marketing image (FMI) sitagliptin/metformin 50 mg/500 mg fixed-dose combination (FDC) tablet with 240 ml water on Day 1 of the relevant treatment period (SitMet850 FDC) after fasting for at least 10 hours.
Drug: Co-administration of 50 mg sitagliptin and 850 mg metformin — Co-administration of 50 mg sitagliptin and 850 mg China sourced metformin as individual tablets with 240 ml water on Day 1 of the relevant treatment period (Sit + Met850) after fasting for at least 10 hours.
Drug: sitagliptin/metformin 50 mg/850 mg tablet — Single dose administration of the FMI sitagliptin/metformin 50 mg/850 mg FDC tablet with 240 ml water on Day 1 of the relevant treatment period (SitMet850 FDC) after fasting for at least 10 hours.

SUMMARY:
This study will test the hypothesis that the Final Market Image (FMI) sitagliptin/metformin 50 mg/500 mg and 50 mg/850 mg (Fixed Dose Combination) FDC tablet and co-administration of corresponding doses of sitagliptin and China-sourced metformin as individual tablets will be bioequivalent based on assessment of the AUC(0-t) and Cmax, for both sitagliptin and metformin.

ELIGIBILITY:
Inclusion Criteria:

* Subject is of Chinese descent
* Subject is in good health
* Subject is a non-smoker

Exclusion Criteria:

* Subject has a history of stroke or chronic seizures
* Subject has a history of cancer
* Subject has had major surgery, donated blood or participated in another investigational study within the past 4 weeks

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 28 participants were randomized in four treatment sequences. Participants had a 7 day minimum washout period between treatments.
Period: Treatment Period 1
Arm/Group | 1. Sit + Met500 / SitMet500 FDC / SitMet850 FDC / Sit + Met850 | 2. SitMet500 FDC / Sit + Met850 / Sit + Met500 / SitMet850 FDC | 3. Sit + Met850 / SitMet850 FDC / SitMet500 FDC / Sit + Met500 | 4. SitMet850 FDC / Sit + Met500 / Sit + Met850 / SitMet500 FDC
Started | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | 1. Sit + Met500 / SitMet500 FDC / SitMet850 FDC / Sit + Met850 | 2. SitMet500 FDC / Sit + Met850 / Sit + Met500 / SitMet850 FDC | 3. Sit + Met850 / SitMet850 FDC / SitMet500 FDC / Sit + Met500 | 4. SitMet850 FDC / Sit + Met500 / Sit + Met850 / SitMet500 FDC
Started | 7 | 7 | 6 (After period 1, one participant was discontinued by the investigator due to a protocol deviation.) | 7
Completed | 7 | 7 | 6 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | 1. Sit + Met500 / SitMet500 FDC / SitMet850 FDC / Sit + Met850 | 2. SitMet500 FDC / Sit + Met850 / Sit + Met500 / SitMet850 FDC | 3. Sit + Met850 / SitMet850 FDC / SitMet500 FDC / Sit + Met500 | 4. SitMet850 FDC / Sit + Met500 / Sit + Met850 / SitMet500 FDC
Started | 7 | 7 | 6 | 7
Completed | 7 | 7 | 6 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 4
Arm/Group | 1. Sit + Met500 / SitMet500 FDC / SitMet850 FDC / Sit + Met850 | 2. SitMet500 FDC / Sit + Met850 / Sit + Met500 / SitMet850 FDC | 3. Sit + Met850 / SitMet850 FDC / SitMet500 FDC / Sit + Met500 | 4. SitMet850 FDC / Sit + Met500 / Sit + Met850 / SitMet500 FDC
Started | 7 | 7 | 6 | 7
Completed | 7 | 7 | 6 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.6 (5.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 28
Region of Enrollment [Number; unit: participants]
  China | 28
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 22 (1.22)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC(0-t)) for Sitagliptin
Description: AUC (0-t) is the area under the curve for the plot showing plasma concentration against time from time zero to the time of the last quantifiable concentration for sitagliptin 50 mg, metformin 500 mg and metformin 850 mg.
Time Frame: baseline through 72 hours postdose
Population: Per-Protocol (PP) set: Participants who completed the study according to the protocol. One participant who discontinued after Treatment Period 1 was not included in the analysis.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Groups:
- Sit 50 mg + Met 500 mg: Participants co-administered 50 mg sitagliptin and 500 mg metformin as individual tablets from all treatment sequences.
- SitMet 50mg/500mg FDC: Participants administered the sitagliptin/metformin 50 mg/500 mg FDC tablet from all treatment sequences.
- Sit 50 mg + Met 850 mg: Participants co-administered 50 mg sitagliptin and 850mg metformin as individual tablets from all treatment sequences.
- SitMet 50mg/850mg FDC: Participants administered sitagliptin/metformin 50 mg/850 mg FDC tablet from all treatment sequences.
Arm/Group | Sit 50 mg + Met 500 mg | SitMet 50mg/500mg FDC | Sit 50 mg + Met 850 mg | SitMet 50mg/850mg FDC
Number analyzed (Participants) | 27 | 27 | 27 | 27
hr*ng/mL
  sitagliptin 50 mg | 1570 (217.40) | 1590 (186.58) | 1520 (228.83) | 1600 (195.05)
  metformin 500 mg | 8350 (1881.70) | 8750 (1920.45) | NA (NA) — Metformin 500 mg was not administered during this treatment. | NA (NA) — Metformin 500 mg was not administered during this treatment.
  metformin 850 mg | NA (NA) — Metformin 850 mg was not administered during this treatment. | NA (NA) — Metformin 850 mg was not administered during this treatment. | 11800 (2849.36) | 13100 (2987.28)

2. Primary Outcome: Cmax for Sitagliptin and Metformin
Description: Cmax is the peak serum concentration of a therapeutic drug after administration; and is used to determine the rate and extent of drug absorption. Cmax is reported for sitagliptin 50 mg, metformin 500 mg and metformin 850 mg.
Time Frame: baseline through 72 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sit 50 mg + Met 500 mg | SitMet 50mg/500mg FDC | Sit 50 mg + Met 850 mg | SitMet 50mg/850mg FDC
Number analyzed (Participants) | 27 | 27 | 27 | 27
ng/mL
  sitagliptin 50 mg | 189 (37.76) | 182 (38.71) | 187 (40.31) | 194 (32.67)
  Metformin 500 mg | 1210 (323.83) | 1310 (383.57) | NA (NA) — Metformin 500 mg was not administered during this treatment. | NA (NA) — Metformin 500 mg was not administered during this treatment.
  Metformin 850 mg | NA (NA) — Metformin 850 mg was not administered during this treatment. | NA (NA) — Metformin 850 mg was not administered during this treatment. | 1790 (488.51) | 1970 (482.69)

ADVERSE EVENTS:
Groups:
- Sit 50 mg + Met 500 mg: AEs reported in participants after co-administration of 50 mg sitagliptin and 500 mg metformin.
- Sit/Met 50 mg/500 mg FDC: AEs reported in participants after administration of the sitagliptin/metformin 50 mg/500 mg fixed dose combination (FDC) tablet.
- Sit 50 mg + Met 850 mg: AEs reported in participants after co-administration of 50 mg sitagliptin and 850 mg metformin.
- Sit/Met 50 mg/850 mg FDC: AEs reported in participants after administration of sitagliptin 50 mg/metformin 850 mg FDC tablet.
Arm/Group | Sit 50 mg + Met 500 mg | Sit/Met 50 mg/500 mg FDC | Sit 50 mg + Met 850 mg | Sit/Met 50 mg/850 mg FDC
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 4/28 | 3/28 | 4/28 | 2/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sit 50 mg + Met 500 mg (N=28) | Sit/Met 50 mg/500 mg FDC (N=28) | Sit 50 mg + Met 850 mg (N=28) | Sit/Met 50 mg/850 mg FDC (N=28)
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 1 | 0
Fever (General disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Leucocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 — Laboratory finding

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. SPONSOR review can be expedited to meet publication guidelines.